CLINICAL TRIAL: NCT06420128
Title: Collaborative Practice in Primary Care: a Comparison of the Global Rate of Potentially Avoidable Hospitalization, Depending on Whether Their General Practitioner is Part of a Primary Care Team. A Cohort Study With a 36-month Follow-up.
Brief Title: Interprofessional Collaborative Practice in Primary Care: Potentially Avoidable Hospitalization
Acronym: SCOPE HPE
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC21_0307
Record Dates: First submitted 2024-05-03; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Hospitalization; Aged; Primary Health Care
Keywords: Collaborative practice; Seniors; Potentially avoidable hospitalization; Primary Care Team

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary care team: Patients whose general practitioner is a member of a primary care team since at least 12 months
  Interventions: Other: Primary care team
- Traditional: Patients whose general practitioner is not part of a primary care team

INTERVENTIONS:
Other: Primary care team — Patients whose general practitioner is a member of a primary care team since at least 12 months
  Groups: Primary care team

SUMMARY:
The World Health Organization supports collaborative practice in primary care, defining it as "when multiple health professionals from different professional backgrounds work together with patients, families, carers and communities to deliver the highest quality of care across settings" (1). Previous research have shown that collaborative practice in primary care improves care pathways, efficiency of care (2,3), job satisfaction among health professionals (4-6), and economic efficiency (3,7). Riverin et al. found a reduction in post-hospitalization mortality with collaborative practice (8).

In France, the establishment of primary care teams following the American model of Centered Medical Homes is encouraged. In the Pays de la Loire region, two models exist: A national and a regional model.

A major issue for patient care team is the care of seniors (9,10).Hospitalizations can have adverse health effects for this population (11,12). 45% of emergency admissions follow by a hospitalization concern them (13).

The hypothesis of the study is that collaborative practice could reduce the global rate of potential avoidable hospitalizations among seniors.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 75 years old and over 65 years old with chronic disease(s), with a general practitioner in Pays de la Loire, affiliated with the general health insurance system and have had at least one healthcare encounter, and residing in the Pays de la Loire region.

Exclusion Criteria:

* Patients whose general practitioner has ceased their practice or changed their affiliation, as well as patients who have switched to a new general practitioner.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Seniors
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of Global rate of potentially avoidable hospitalization | 36 months
  Comparison of the global rate of potentially avoidable hospitalization of seniors, depending on whether their general practitioner is a member of a primary care team. Use of reimbursement data of Health Insurance System.

SECONDARY OUTCOMES:
Comparison of criterion of quality | 36 months
  Comparison of criterion of quality (rate of potentially avoidable hospitalization with emergency enter, rate of potentially avoidable hospitalization for patients with chronic disease(s), rate of rehospitalization at one month, mortality in post-hospitalization and rate of emergency admission), depending on whether their general practitioner is a member of a primary care team. Use of reimbursement data of Health Insurance System.
Comparison of Global rate of potentially avoidable hospitalization depending the model of primary care team | 36 months
  Comparison of Global rate of potentially avoidable hospitalization depending the model of primary care team Description: comparison of global rate of potentially avoidable hospitalization depending general practitioner is a member of a national model of primary care team or a regional model of primary care team. Use of reimbursement data of Health Insurance System.
Medico-economic evaluation | 36 months
  To determine health expenditures per patient, annual and total. Use of reimbursement data of Health Insurance System.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No